CLINICAL TRIAL: NCT03491813
Title: Comparison Between Centrally Measured Blood Pressure and Automated Blood Pressure Monitoring for Detection of Early Kidney Dysfunction in Patients With Primary Hypertension
Brief Title: Comparisonbetween Primary Hypertension Monitoring Methods for Detection of Early Kidney Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nader Nabil, Principal Investigator, Assiut University
Other Study IDs: Hypertension and CKD
Record Dates: First submitted 2018-03-19; First posted 2018-04-09 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Primary Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: oscillometric device — The blood pressure will be measured by the Automatic blood pressure monitor(Oscillometric) named the OMRON M2 basic® device was provided by Omron Healthcare company.
  This monitor uses inflation by Fuzzy-Logic controlled by electric pump and an automatic rapid pressure release valve for the deflation , its cuff allows BP measurements in arm circumference of 22-42 cm. The device measure BP and pulse rate with a pressure range of 0-299 mmHg and pulse rate range of 40-180 beats/min.

SUMMARY:
The present study aims to show the difference of blood pressure monitored centrally and automated BP monitoring among patients with primary hypertension for early detection of kidney dysfunction

DETAILED DESCRIPTION:
Hypertension is well known as the silent killer, There is a close relationship between blood pressure levels and the risk of cardiovascular events, strokes and kidney disease.

Diabetes and hypertension cause up to two-thirds of chronic kidney disease , chronic kidney disease is a common condition characterized by evidence of kidney damage or dysfunction.

chronic kidney disease is currently classified based on a patient's estimated glomerular filtration rate and urinary albumin excretion rate , clinicians look for markers of renal damage (e.g., abnormalities of urinary sediment or organ structure) to diagnose chronic kidney disease in people with estimated glomerular filtration rate of <60 mL/min/1.73 m2.

Age distribution for hypertension showed progressive rise in blood pressure with increasing age. Age-related hypertension appears to be predominantly systolic rather than diastolic. The third NHANES survey reported that the prevalence of hypertension grows significantly with increasing age in all sex and race groups. In another study, the incidence of hypertension appeared to increase approximately 5% for each 10-year interval of age Because Central blood pressure is considered better than peripheral blood pressure in predicting cardiovascular events, due to wave reflections and viscoelastic properties of the arterial wall Now a day several non-mercury techniques have been developed during the last ten years in order to gradually supplant the mercury-auscultatory method, such as the automatic electronic devices using algorithms based on the oscillometric technique.

Over the last ten years , different protocols are used to validate the accuracy of blood pressure measuring devices , several automated devices have been successfully validated using established protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 Years to 70 Years old .
2. Patients who have history of primary hypertension either on medical treatment or not .

Exclusion Criteria:

1. All patients with 2ry hypertension.
2. Diabetic patients.
3. Patients with ESRD on regular dialysis .
4. Patients with creatinineclearance >30ml/min .
5. collagen diseases

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with primary hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Detection of kidney dysfunction in patients with primary hypertension | 1 year
  Detection of kidney dysfunction by estimation of creatinine clearance using crclcockroftـGault equation.
  In patients with primary hypertension and blood pressure will measured by two methods
  1. Central Blood Pressure monitoring through non-invasively using a new well calibrated device named Mobil-O- Graph .( Cuff-based oscillometry at the brachial artery)
  2. Automatic blood pressure monitor (Oscillometric) named the OMRON M2 basic® device was provided by Omron Healthcare company.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdel Galeel, MD, Study Chair — Assiut University; Doaa Fouad, Study Director — Assiut University

REFERENCES:
- [Background] Cornoni-Huntley J, LaCroix AZ, Havlik RJ. Race and sex differentials in the impact of hypertension in the United States. The National Health and Nutrition Examination Survey I Epidemiologic Follow-up Study. Arch Intern Med. 1989 Apr;149(4):780-8. PMID 2784957
- [Background] Burt VL, Whelton P, Roccella EJ, Brown C, Cutler JA, Higgins M, Horan MJ, Labarthe D. Prevalence of hypertension in the US adult population. Results from the Third National Health and Nutrition Examination Survey, 1988-1991. Hypertension. 1995 Mar;25(3):305-13. doi: 10.1161/01.hyp.25.3.305. PMID 7875754
- [Background] Pickering T. The case for a hybrid sphygmomanometer. Blood Press Monit. 2001 Aug;6(4):177-9. doi: 10.1097/00126097-200108000-00002. PMID 11805464